CLINICAL TRIAL: NCT04978259
Title: Long-term Follow-up of a Randomized Multicenter Trial on Impact of Long-COVID in Hospitalized COVID-19 Patients
Brief Title: SOLIDARITY Finland Long-COVID (Remdesivir Long-term Follow-up Study of COVID Patients)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinical Urology and Epidemiology Working Group (Other Government)
Collaborators: University of Helsinki (Other); World Health Organization (Other); Helsinki University Central Hospital (Other); Hyvinkää Hospital (Other); Kanta-Häme Central Hospital (Other Government); Kuopio University Hospital (Other); Oulu University Hospital (Other); Porvoo Hospital (Unknown); Seinajoki Central Hospital (Other); Mikkeli Central Hospital (Other); Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Kari Tikkinen, Professor, Clinical Urology and Epidemiology Working Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOL21
Record Dates: First submitted 2021-07-20; First posted 2021-07-27 (Actual); Last update posted 2022-07-15 (Actual); Status verified 2022-06

CONDITIONS: Covid19
Keywords: long-COVID; COVID; randomised trial; evidence-based medicine; remdesivir; symptoms; quality of life; mortality; morbidity; genetics; Covid19
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome | interventions — remdesivir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care plus remdesivir (Experimental): Local standard of care plus daily remdesivir infusion for up to 10 days (or until discharge)
  Interventions: Drug: Remdesivir
- Standard of care (No Intervention): Local standard of care

INTERVENTIONS:
Drug: Remdesivir — Intravenous remdesivir during hospital stay up to 10 days in addition to standard care.
  Arms: Standard of care plus remdesivir

SUMMARY:
SOLIDARITY Finland Long-COVID trial assesses the effects of remdesivir + standard of care (SoC) vs. only SoC on long-COVID symptoms and quality of life (QoL) using questionnaires at one and two years post-discharge.

Objectives i) Long-COVID symptoms

* To investigate the effect of remdesivir (vs. SoC) on the occurrence of symptoms that have been associated with the long-COVID syndrome. The questionnaires will take place 1 and 2 years after the hospital admission.
* The symptom questionnaire - that will be completed by patients at one and two years - measures basic patient information (age, height, weight, smoking status, major comorbidity, and working status) and a wide variety of potential long-COVID-symptoms and their bother (1. Fatigue; 2. Attention deficits; 3. Memory problems; 4. Sleeping difficulties; 5. Depressive mood; 6. Anxiety; 7. Dizziness; 8. Headache; 9. Tinnitus; 10. Paresthesias; 11. Changes in taste/smell perceptions; 12. Postexertional malaise; 13. Palpitations; 14. Chest discomfort; 15. Nausea; 16. Skin rash; 17. Joint aches; 18. Muscle pains; 19. Continuous cough; 20. Respiratory tract mucous discharges) in remdesivir and usual care arms

ii) Quality of life

* EQ-VAS: to compare patients' quality of life in remdesivir and usual care arms.
* EQ-5D-5L questionnaire assesses the following domains: 1. Mobility; 2. Self-care; 3. Usual activities; 4. Pain and discomfort; 5. Anxiety and depression; 6. The VAS of subjective perception of overall health.

Additionally (at 1 or 2 years; depending on future funding and ethical approval decisions; currently the study has ethical approval for long-COVID and quality of life assessments only):

* The Finnish healthcare registries (Statistics Finland Mortality Database and the HILMO Care Register for Health Care) will be used to estimate long-term mortality and incidence of major comorbidity in remdesivir and usual care arms
* Lung function will be assessed using spirometry and diffusing capacity, as well as the six-minute walk test (6 mwt) in remdesivir and usual care arms
* Whole-genome genotyping will be performed for a genome-wide association study to investigate genetic correlates of long-COVID-19 -symptoms in remdesivir and usual care arms

UPDATE 02.02.2022:

Primary outcomes will comprise the following:

1. EQ-VAS
2. EQ-5D-5L, summary
3. Does the patient feel recovered from COVID-19-infection at one year or not? (question no. 10)
4. Fatigue (questionnaire, question no. 14)
5. Exertional dyspnea (question no. 12)

DETAILED DESCRIPTION:
The SOLIDARITY Finland Long-COVID is the long-term follow-up of the remdesivir sub-study of the SOLIDARITY Finland. (Following the WHO core protocol with local adjustments, the SOLIDARITY Finland is an adaptive, randomized, open-label clinical trial evaluating the safety and efficacy of possible therapeutic agents in hospitalized adult patients diagnosed with COVID-19.)

Study population Adult patients with confirmed SARS-2-CoV-2 admitted to the hospital ward or the intensive care unit (ICU) were included. Adult hospital patients, with definite COVID-19 and, as per the responsible doctor, no contraindication to the study drugs were entered into the online electronic data collection system and randomly allocated between the local standard of care alone or local standard of care plus remdesivir (daily infusion until discharge or up to ten days). Between July 2020 and January 2021, 208 patients were recruited from 13 hospitals, of which 114 were randomized to receive remdesivir plus usual care and 94 to receive usual care only. (These patients (if alive; n=202 or less) will be invited to participate in the SOLIDARITY Finland Long-COVID.) During patient recruitment at the hospital phase of the study, the following data was collected: 1) hospital and randomizing doctor; 2) confirmation that patient has provided consent, 3) patient identifiers, age, and sex, 4) major comorbidities, 5) COVID severity.

Consent:

All patients have already consented to SOLIDARITY Finland (in-hospital study). In the SOLIDARITY Finland Long-COVID, patients will receive, by mail, an information letter, consent form, and questionnaires. The mail will be sent three days before the anniversary of the randomization day during hospitalisation. They may reply by i) sending back the completed documents, ii) scheduling a phone call with an investigator for an interview, or iii) declining participation. If the patient does not reply in 14 days (from the day the investigators sent the questionnaire to the patient), the investigators will send one reminder by mail and, if there will not be a reply, then the investigators will approach the patient via telephone at around 10 days from the reminder mail. The phone call will be attempted twice: during and after office hours. If the patient will not answer the phone, the investigators will also send a text message to inform them about the reason for our attempted phone call.

Questionnaire (symptoms and characteristics):

Our multidisciplinary team of clinicians, methodologists, and patient partners developed a questionnaire that records basic patient information. This will include i) date of completing the questionnaire, ii) age, iii) height and weight, iv) smoking status (never, ex-smoker, current smoker), v) possible comorbidities, and whether diagnosed before or after COVID-19-infection (obstructive sleep apnea, stroke, coronary artery disease, diabetes, hypertension, cancer, and any psychiatric disease), vi) employment (student, unemployed, employed, sickness allowance, retired), vii) working capability in comparison to the pre-COVID-19 state, viii) physician visits due to symptoms associated with COVID-19, ix) physician-diagnosed long-COVID-19 syndrome. Questionnaires will also document long-term symptoms. Relevant long-COVID-19 -symptoms (in total 20) were identified from recent publications and review articles. This same questionnaire will be used at one and two years. Exertional and cardiopulmonary symptoms potentially related to COVID include fatigue, postexertional malaise, dyspnea during exercise, chest discomfort, palpitations, cough, and respiratory mucous discharges. Main neuropsychiatric symptoms potentially related to COVID include generalized fatigue, attention and memory deficits, sleeping difficulties, depression and anxiety, dizziness, and even sensory disturbances such as paresthesias and changes in taste or smell perceptions. Other commonly encountered symptoms potentially related to COVID include widespread pains (muscle and joint pains, headache), skin rash, nausea, and fever. The burden from each individual symptom is an ordinal variable and will be graded from 0 to 3, where 0 represents no symptom, 1 represents mild bother, 2 moderate bother, and 3 severe bother due to the symptom. Dyspnea is assessed in accordance with the Modified Medical research council dyspnea scale (mMRC) from 0 to 4, where 0 represents dyspnea only with strenuous exercise, and 4 the presence of dyspnea even with mild physical activity, e.g., dressing clothes. To capture the dimensions of recovery, the investigators will use the Core Outcome Measure for Recovery, which has been recommended for use in COVID-19 research.

Quality of life:

The investigators have obtained permission from EuroQol to use the EQ-5D-5L questionnaire to record the patient's QoL. EQ-5D-5L assesses the domains of mobility, self-care, usual daily activities, general pain/discomfort, anxiety/depressions, and an overall impression of health. The first five domains are graded from 1 to 5, while the last uses the visual analogue scale from 0 to 100. Due to our multiethnic patient population, the questionnaires have been translated in the following languages: Albanian, Arabic, English, Estonian, Farsi, Finnish, Russian, Somali, and Swedish. The above-mentioned questionnaire (Finnish language version as the original) has also been translated into these languages.

Data security and future use of data:

Patient information will be encrypted and held securely by the Sponsor. Those analyzing it will use only pseudonymized data, and no identifiable patient details will appear in publications. Data from questionnaires will also be analyzed using pseudonymized data. The investigators have taken care to limit the questions to necessary and clinically relevant aspects related to long-COVID.

UPDATE 02.02.2022:

Primary outcomes will comprise the following:

1. EQ-VAS
2. EQ-5D-5L, summary
3. Does the patient feel recovered from COVID-19-infection at one year or not? (question no. 10)
4. Fatigue (questionnaire, question no. 14)
5. Exertional dyspnea (question no. 12)

To avoid problems related to multiple testing, the trial analysis will be focused on the five most relevant outcomes (listed above). This decision was done before examining the accumulated data, and by consulting statistical experts neither who had seen study data.

Variables collected via questionnaire:

i) Symptoms: 20 symptoms are measured as follows; each range from 0 to 3 (0 = No symptom. 1 = Symptom exists and causes small bother. 2 = Symptom exists and causes moderate bother. 3 = Symptom exists and causes severe bother.) ii) QoL: Using the EQ-VAS and EQ-5D-5L to compare domain-specific scores between the two treatment arms.

Additional variables (at 1 or 2 years; depending on future funding and ethical approval decisions; currently the study has ethical approval for long-COVID and quality of life assessments only):

* Registry data: (UPDATE 02.02.2022) Mortality data with dates are obtained from Digital and Population Data Services Agency during early spring 2022. Later, underlying causes of death will be obtained from Statistics Finland and classified according to the International Statistical Classification of Diseases and Related Health Problems, 10th revision). In line with the Finnish regulations, any consent will not be required from the study patients to acquire information on their census data, vital status, and causes of death for registry research purposes. Comorbidity will be obtained from Finnish Institute for Health and Welfare THL. These will be performed through linkage the patient national identification number to registry records. This study is unlikely well-powered to measure changes in mortality; however, being aware of the vital status is important for the overall follow-up of study participants.
* Lung tests are also planned. Spirometry parameters are continuous variables as absolute values (liters = L; liters per second = L/s), percentage of reference values, and z-values. These include VC, FVC, FEV1, FEV1/VC, peak expiratory flow (PEF), the maximal expiratory flow at 50 % (MEF50), and the forced expiratory time (FET). Spirometry will be performed with a bronchodilator test to assess the changes between baseline and after bronchodilation. Diffusing capacity parameter DLCO is a continuous variable with ml/min/mmHg as the unit.
* Genome sequence analyses are also planned to identify potential single-nucleotide polymorphisms that would associate with long-COVID symptoms and the effect of remdesivir.

Subgroup analyses:

For the primary outcomes, a priori planned subgroup analysis will be performed for whether the patient needed oxygenation at hospital admission (the investigators hypothesize that the treatment effect is larger for those without extra oxygen than those with extra oxygen at hospital admission).

Comparisons between the two treatment arms will be performed as follows:

* Descriptive statistics: Descriptive statistics will be presented with numbers and percentages for categorical variables and means, standard deviation, and range for continuous variables. In the case of clearly skewed continuous variables, they will be presented with median, interquartile range (25th and 75th percentiles), and range. Demographics and baseline characteristics will be presented with descriptive statistics without any hypothesis testing.
* Continuous variables will be subject to repeated measures mixed models or appropriate non-parametric alternatives.
* Binary response variables will be analyzed using logistic regression (possibly adjusting for within-subject dependencies by generalized estimating equations or mixed models) or chi-square/Mantel-Haenszel tests.
* If missing data is regarded as having a significant effect on the conclusions of the trial, sensitivity analyses with different methods for handling missing data will be included. The differences between respondents and non-respondents will be assessed using available baseline variables.

Statistical analyses in more detail:

1. EQ-VAS

   * Mann-Whitney test, when the treatment arm is the only variable.
   * Regression analysis to adjust possible imbalances. Linear regression, if VAS scores are not concentrated around either extreme of the scale.
2. EQ-5D-5L, summary.

   - Proportions of respondents in both groups by categories (Mobility, Self-Care, Usual Activities, Pain/Discomfort, Anxiety/Depression).
3. Does the patient feel recovered from COVID-19-infection at one year or not? (question no. 10)
4. Fatigue (questionnaire, question no. 14)

   - Logistic regression analysis. "No symptom" and "Mild symptoms" will be analyzed together against "Moderate symptoms" and "Severe symptoms".
5. Exertional dyspnea (question no. 12) - Logistic regression analysis. mMRC categories 0 and 1 will be analyzed together against categories 2-4.

ELIGIBILITY:
Inclusion Criteria:

* Alive patients who attended the SOLIDARITY Finland remdesivir sub-study

Eligibility criteria for SOLIDARITY Finland remdesivir -study:

Inclusion criteria:

* Adult patients, 18 years and older
* Laboratory-confirmed SARS-CoV-2 infection
* Admitted to the hospital ward or the intensive care unit (ICU)
* Patient provides written informed consent prior to initiation of the study OR close relative/legal representative provides written informed consent prior to initiation of the study according to the presumed will of the patient when patient is unable to give consent.
* No anticipated transfer within 72 hours to a non-study hospital

Exclusion Criteria:

* Severe co-morbidity with life expectancy <3 months according to investigators assessment
* ASAT/ALAT > 5 times the upper limit of normal
* Acute co-morbidity within 7 days before inclusion such as myocardial infarction or unstable angina pectoris (not including troponin elevation due to infection)
* Pregnancy or breast feeding
* Any reason why, in the opinion of the investigators, the patient should not participate
* Subject participates in a potentially confounding drug or device trial during the course of the study
* Already receiving the study drug
* Renal failure (eGRF < 30 mL/min) or dialysis/continuous veno-venous hemofiltration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2021-07-24 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
EQ-VAS | 1 year
  EQ-VAS is a patient-reported outcome measure of quality of life on a scale from 0 to 100.
  The minimum scores mean a worse outcome.
EQ-5D-5L | 1 year
  Quality of life measure of five domains, including mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
Recovering from COVID-19 infection | 1 year
  Question: How do you feel you have recovered from the COVID-19 infection you had one year ago? Five options from "fully recovered" to "not recovered at all"
Fatigue | 1 year
  The presence of fatigue as: 0 = no fatigue, 1 = mild fatigue, 2 = moderate fatigue, and 3 = severe fatigue.
Exertional dyspnea | 1 year
  mMRC scale measures the degree of disability that breathlessness poses on everyday activities on a scale from 0 to 4.
Long-COVID symptoms | 1 year
  Infection affected quality of life in the last month as: 0 = No symptoms of infection, 1 = Slight harm, 2 = Moderate harm, 3 = Severe harm

SECONDARY OUTCOMES:
EQ-VAS | 2 year
  EQ-VAS is a patient-reported outcome measure of quality of life on a scale from 0 to 100 The minimum scores mean a worse outcome.
EQ-5D-5L | 2 year
  Quality of life measure of five domains, including mobility, self-care, usual activities, pain/discomfort and anxiety/depression.
Recovering from COVID-19 infection | 2 year
  Question: How do you feel you have recovered from the COVID-19 infection you had one year ago? Five options from "fully recovered" to "not recovered at all"
Fatigue | 2 year
  The presence of fatigue as: 0 = no fatigue, 1 = mild fatigue, 2 = moderate fatigue, and 3 = severe fatigue.
Exertional dyspnea | 2 year
  mMRC scale measures the degree of disability that breathlessness poses on everyday activities on a scale from 0 to 4.
Long-COVID symptoms | 2 year
  Infection affected quality of life in the last month as: 0 = No symptoms of infection, 1 = Slight harm, 2 = Moderate harm, 3 = Severe harm

OTHER OUTCOMES:
Mortality | Long-term at one year
  Obtiained from health care registries
Incidence of comorbidity | Long-term at one year, obtained from registries
  Obtiained from health care registries
Lung function | 2 years post-discharge
  Spirometry: VC, FVC, FEV1, FEV1/VC, peak expiratory flow (PEF), the maximal expiratory flow at 50 % (MEF50), and the forced expiratory time (FET)
Lung function | 2 years post-discharge
  Lung diffusion capacity: Diffusing capacity parameter DLCO is a continuous variable with ml/min/mmHg as the unit.
Lung function | 2 years post-discharge
  6-minute walking test
Whole-genome sequencing | 2 years post-discharge

CONTACTS AND LOCATIONS:
Overall Officials: Kari AO Tikkinen, MD PhD, Study Director — University of Helsinki; Olli Nevalainen, MD PhD, Principal Investigator — University of Helsinki
Locations (1):
- University of Helsinki, Helsinki, Finland

REFERENCES:
- [Derived] Grundeis F, Ansems K, Dahms K, Thieme V, Metzendorf MI, Skoetz N, Benstoem C, Mikolajewska A, Griesel M, Fichtner F, Stegemann M. Remdesivir for the treatment of COVID-19. Cochrane Database Syst Rev. 2023 Jan 25;1(1):CD014962. doi: 10.1002/14651858.CD014962.pub2. PMID 36695483

DOCUMENTS (1):
  • Informed Consent Form (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/59/NCT04978259/ICF_001.pdf